CLINICAL TRIAL: NCT02808078
Title: Visually-guided Gait Training in Paretic Patients During First Rehabilitation: a Randomized Controlled Trial
Brief Title: Gait Adaptation for Stroke Patients With Augmented Reality
Acronym: GASPAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philippe Terrier (Network)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, Philippe Terrier, Senior Researcher, Clinique Romande de Readaptation
Organization: Clinique Romande de Readaptation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CliniqueRR-04
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Traumatic Brain Injury; Spinal Cord Injury
Keywords: Instrumented treadmill; Augmented reality; Neurorehabilitation; Gait disorders
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Spinal Cord Injuries; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmented reality training (Experimental): Gait training with augmented reality
  Interventions: Device: Gait training with augmented reality
- Standard training (Active Comparator): Gait training without augmented reality
  Interventions: Device: Standard training

INTERVENTIONS:
Device: Gait training with augmented reality — 20 sessions (30 min. duration) over 4 weeks of gait training with augmented reality.
  Arms: Augmented reality training
Device: Standard training — 20 sessions (30 min. duration) over 4 weeks of gait training without augmented reality.
  Arms: Standard training

SUMMARY:
The GASPAR trial is a pragmatic, parallel-arms, single-center, non-blinded, superiority randomized control trial in neurorehabilitation. The main objective is to test whether a 4 weeks gait rehabilitation program that uses augmented reality is superior to a conventional treadmill training program of equivalent intensity. Baseline assessments precede allocation, which consists in blocking randomization (2:1 ratio) with stratification according to the disease etiology. Post-intervention assessments serve to compare the short-term efficacy of the intervention between the two groups. Three months after discharge, follow-up assessments take place to detect potential long-term effects.

DETAILED DESCRIPTION:
After a lesion to the central nervous system, many patients suffer from a diminished walking capability. During the first rehabilitation phase, specific cares help the recovery of motor function to offer the best chances of returning to normal walk. For example, the repeated practice of walking exercises facilitates the gain of muscular strength and stimulates motor relearning. However, in patients, who have finished the first rehabilitation phase, it is often observed strong limping, unsteady gait, and a bad management of obstacle clearance. Thus, these individuals fall frequently, with risk of severe injury. The aim of the study is to assess the efficacy of gait training on a treadmill equipped with an augmented reality system. Shapes are displayed onto the treadmill belt with a projector (beamer): the patient adapts his/her gait to the drawing that unfolds in front of him/her. It is possible to train gait symmetry for coordination enhancement or to exercise obstacle clearance and gait agility. Another advantage of this type of treadmill is the capability to continuously analyze gait with integrated sensors and, hence, to give real-time feedback to the patient. Whereas the method seems promising, thorough studies that would confirm its efficacy are lacking. Therefore, the investigators seek to conduct a randomized controlled trial to compare visually-guided gait training with a more classical training method. During four weeks, participants will train, according to their abilities, three to five times a week during 30 minutes on the augmented-reality treadmill. A group of control patients will train at comparable intensity but without the visual guidance of gait. Using the data collected during the training sessions, the investigators will study whether the evolution of locomotor function differs between both groups. Furthermore, several questionnaires will be filled in by the participants to document the self-evaluation of their progress. In the long term, the investigators expect to first improve the efficacy of gait rehabilitation and second to better understand the recovery process of locomotor function during the first months after a stroke.

ELIGIBILITY:
Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Informed Consent as documented by signature
* Stroke patients, patients with traumatic brain injury, or patients with spinal cord injury in the acute to sub-acute phase (maximum 40 days after the incident)
* Need for gait rehabilitation in reason of at least one of the following conditions: Paresis of the lower extremities. Severe balance disorders. No walking at entry due to the neurological injury
* Ability to walk 2 minutes without or with minimal aid, namely: With the help of one person, or: With walking aid (cane, walker)

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Age < 18 years
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.) that may threaten the health in case of sustained exercise.
* Concomitant gait disorders induced by acute to sub-acute musculoskeletal injuries, e.g. fracture of the lower extremities.
* Severe pre-existent gait disorders that deeply affect walking abilities and gait pattern, either due to musculoskeletal (e.g. severe osteoarthritis) or neurological (e.g. Parkinson's disease) etiologies.
* Severe non-corrected visual impairment
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | Pre-intervention (week 0), Post-intervention (week 5)
  Walking speed, measured with the 2-minute walk test

SECONDARY OUTCOMES:
Change in postural control | Pre-intervention (week 0), Post-intervention (week 5)
  Capabilities to ensure an optimal postural control. Measured with the Berg Balance test
Fear of falling during the hospitalization | week 5
  Subjective assessment of the fear of falling. Measured with the adapted Falls Efficacy Scale (FES)
Fear of falling at home | after discharge at 3-4 month
  Subjective assessment of the fear of falling. Measured with the adapted Falls Efficacy Scale (FES)
Quality of life at home | after discharge at 3-4 month
  Short-Form 36 questionnaire (SF-36)
Perception of the intervention | During the intervention, week 2 and 4
  purpose-designed questionnaire that will ask to the participant about their perception of the intervention. The questionnaire will evaluate the satisfaction with intensity, duration and difficulty of the intervention. Other questions will ask about the perceived training effects on walking speed and confidence.
Changes in stride and step lengths | In every gait training sessions, from week 1 to week 4
  Measured with the embedded sensors of the treadmills
Changes in stride and step durations | In every gait training sessions, from week 1 to week 4
  Measured with the embedded sensors of the treadmills
Change in step width | In every gait training sessions, from week 1 to week 4
  Measured with the embedded sensors of the treadmills
Change in left/right asymmetry of step lengths | In every gait training sessions, from week 1 to week 4
  Measured with the embedded sensors of the treadmills
Change in left/right asymmetry of step durations | In every gait training sessions, from week 1 to week 4
  Measured with the embedded sensors of the treadmills
Changes in stance and swing phases | In every gait training sessions, from week 1 to week 4
  Measured with the embedded sensors of the treadmills
Change in gait variability | In every gait training sessions, from week 1 to week 4
  Stride-to-stride variability of gait parameters (outcomes 7-12)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Terrier, PhD, Principal Investigator — Institute for Research in Rehabilitation and Clinique romande de réadaptation
Locations (1):
- Clinique Romande de Réadaptation, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, final anonymized database will be made available through a specialized online repository

REFERENCES:
- [Derived] Rossano C, Terrier P. Visually-guided gait training in paretic patients during the first rehabilitation phase: study protocol for a randomized controlled trial. Trials. 2016 Oct 27;17(1):523. doi: 10.1186/s13063-016-1630-8. PMID 27788679